CLINICAL TRIAL: NCT04619264
Title: Impact of Minimally Invasive Restorative Techniques on Pregnant Women Oral Health Related Quality of Life: a Randomized Clinical Trial
Brief Title: Impact of Minimally Invasive Restorative Techniques on Pregnant Women Oral Health Related Quality of Life
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: minimally invasive & OHRQoL
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Quality of Life; Dental Caries
Keywords: Minimally Invasive Caries Removal; Oral Health Related Quality of Life
MeSH Terms: conditions — Dental Caries | interventions — Papacarie; Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Papacarie-Duo (Experimental)
  Interventions: Drug: Papacarie
- Atraumatic Restorative Treatment (Active Comparator)
  Interventions: Procedure: Atraumatic Restorative Treatment

INTERVENTIONS:
Drug: Papacarie — First, tooth was cleaned with a wet cotton pellet. The gel was inserted using disposable syringe tip into the cavity and its color changed from clear to cloudy indicating the presence of infected tissues. After 40 seconds, the softened carious tissue was removed using excavator by gentle pressure. The remaining gel was removed with a cotton pellet. The procedure was repeated until there was no change in the gel color indicating that there was no more infected tissue.
  Other Names: Papacarie-Duo
  Arms: Papacarie-Duo
Procedure: Atraumatic Restorative Treatment — The tooth was cleaned with a wet cotton pellet to remove debris and plaque and then isolated with cotton rolls to promote a dry environment. Caries was removed using a sharp excavator and the cavity was cleaned using a small wet cotton pellet and dried with a dry cotton pellet.
  Other Names: ART
  Arms: Atraumatic Restorative Treatment

SUMMARY:
Aim of the study was to compare the effect of chemo-mechanical caries removal methods using Papacarie-Duo and alternative restorative treatment (ART) on the Oral Health Related Quality of Life (OHRQoL) of pregnant women.

DETAILED DESCRIPTION:
A randomized controlled clinical trial was conducted in 2019 and included 162 pregnant women visiting family health centers in Alexandria, Egypt with mild to moderate dental pain due to caries. Participants were randomly assigned into Papacarie-Dup group (n=82) and ART group (n=80). The outcome variable was percent change in OHRQoL measured by OHIP-14.

ELIGIBILITY:
Inclusion Criteria:

* Having at least one carious lesion involving dentine with lesion accessible to hand instruments (International Caries Detection and Assessment System score= 5 or 6).
* Suffering from at least mild dental pain as identified by a score of at least 5mm on a Visual Analogue Scale (VAS) 100-mm-long.

Exclusion Criteria:

* Pregnant women with acute pulpitis, swelling or fistula.
* Uncooperative patients and those who refused to participate.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females in the first or second trimester
Enrollment: 162 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Change in Oral Health Related Quality of Life | up to 6 months
  This was assessed by measuring changes between the Oral Health Impact Profile-14 (OHIP-14). The OHIP-14 includes 14 questions in seven dimensions with two questions for each dimension: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. Responses to the OHIP-14 items were measured on a 5-pont Likert scale ranging from never = 0; hardly ever = 1; occasionally = 2; fairly often = 3; to very often = 4. The OHIP-14 score is the sum of the scores of the 14 statements and ranges from 0 to 56 and from 0 to 8 for each dimension with higher scores indicating higher frequency of negative impact.
Retention of the final restoration | up to 6 months
  The scoring system was as follows: 0=present, without defect; 1=present, small defects on the margin measuring less than 0.5 mm in depth, with no need for repair; 2=present, small defects on the margin measuring 0.5 to 1.0 mm in depth, with need for repair; 3=present, gross defects on the margin measuring 1.0 mm or more in depth, with need for repair; 4=absent, restoration completely lost, need for treatment; 5=absent, other treatment had been performed for some reason; 6=tooth absent for some reason; 7=present, wear on surface less than 0.5 mm, with no need for replacement; 8=present, wear on surface greater than 0.5 mm, with need for replacement; 9=diagnosis impossible. Restorations having a score of 0, 1 or 7 were considered successful and those receiving a score of 2, 3, 4 or 8 were considered failures.

CONTACTS AND LOCATIONS:
Overall Officials: May M Adham, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Mona K ElKashlan, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Wafaa E Abdelaziz, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Family Health Centers, Alexandria, Egypt

REFERENCES:
- [Background] Kikwilu EN, Frencken J, Mulder J. Impact of Atraumatic Restorative Treatment (ART) on the treatment profile in pilot government dental clinics in Tanzania. BMC Oral Health. 2009 Jun 8;9:14. doi: 10.1186/1472-6831-9-14. PMID 19505294
- [Background] Matsumoto SF, Motta LJ, Alfaya TA, Guedes CC, Fernandes KP, Bussadori SK. Assessment of chemomechanical removal of carious lesions using Papacarie Duo: randomized longitudinal clinical trial. Indian J Dent Res. 2013 Jul-Aug;24(4):488-92. doi: 10.4103/0970-9290.118393. PMID 24047844
- [Background] Musskopf ML, Milanesi FC, Rocha JMD, Fiorini T, Moreira CHC, Susin C, Rosing CK, Weidlich P, Oppermann RV. Oral health related quality of life among pregnant women: a randomized controlled trial. Braz Oral Res. 2018;32:e002. doi: 10.1590/1807-3107bor-2018.vol32.0002. Epub 2018 Jan 22. PMID 29364329
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Freitas MCCA, Fagundes TC, Modena KCDS, Cardia GS, Navarro MFL. Randomized clinical trial of encapsulated and hand-mixed glass-ionomer ART restorations: one-year follow-up. J Appl Oral Sci. 2018 Jan 18;26:e20170129. doi: 10.1590/1678-7757-2017-0129. PMID 29364343
- [Background] Al Habashneh R, Khader YS, Salameh S. Use of the Arabic version of Oral Health Impact Profile-14 to evaluate the impact of periodontal disease on oral health-related quality of life among Jordanian adults. J Oral Sci. 2012 Mar;54(1):113-20. doi: 10.2334/josnusd.54.113. PMID 22466895
- [Background] Motta LJ, Bussadori SK, Campanelli AP, Silva AL, Alfaya TA, Godoy CH, Navarro MF. Efficacy of Papacarie((R)) in reduction of residual bacteria in deciduous teeth: a randomized, controlled clinical trial. Clinics (Sao Paulo). 2014;69(5):319-22. doi: 10.6061/clinics/2014(05)04. PMID 24838896
- [Derived] Adham MM, El Kashlan MK, Abdelaziz WE, Rashad AS. Comparison of two minimally invasive restorative techniques in improving the oral health-related quality of life of pregnant women: a six months randomized controlled trial. BMC Oral Health. 2021 Apr 30;21(1):221. doi: 10.1186/s12903-021-01581-5. PMID 33931037